CLINICAL TRIAL: NCT00580684
Title: Long-Term Efficacy of Pneumococcal Conjugate 7-Valent Vaccine Versus Plain Polisaccharide Pneumococcus Vacine in Reducing Pneumococcal Nasopharyngeal Carriage of Children.
Brief Title: Study Comparing Prevenar® to Pneumo 23 in Reducing Carriage in Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0887X-101198
Record Dates: First submitted 2007-12-21; First posted 2007-12-27 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Vaccines, Pneumococcal; Vaccines, Pneumococcal Conjugate Vaccine
Keywords: pneumococcus conjugated vaccine 7 valent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G1 (Active Comparator): G1: prevenar
  Interventions: Biological: pneumococcus conjugate vaccine 7 valent to reduce carriage
- G2 (Active Comparator): G2: pneumo 23
  Interventions: Biological: pneumococcus conjugate vaccine 7 valent to reduce carriage

INTERVENTIONS:
Biological: pneumococcus conjugate vaccine 7 valent to reduce carriage — plain polisacaride vaccine 23 valent to reduce carriage

SUMMARY:
To compare the ability of Prevnar® to Pneumo® 23 in reducing and preventing nasopharyngeal carriage of vaccine-type pneumococci one year after respective immunization. To evaluate the rate of penicillin-resistant pneumococci in nasopharyngeal carriage.

DETAILED DESCRIPTION:
This study will require 6 months to be completed (3 months for nasopharyngeal samples collection; 3 months dor analysis). Each child will participate for a 1 day period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children between
* 2 to 9 years old.
* No history of antibiotic use prior 1 month of enrollment
* No history of invasive pneumococcal disease

Ages: 2 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 101 (Actual)
Dates: Start 2003-09; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
To compare the ability of Prevnar® to Pneumo® 23 in reducing and preventing nasopharyngeal carriage of vaccine-type pneumococci one year after respective immunization. | 12 months

SECONDARY OUTCOMES:
To evaluate the rate of penicillin-resistant pneumococci in nasopharyngeal carriage. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer